CLINICAL TRIAL: NCT02951806
Title: Effect of Slow Injection of Fentanyl on the Incidence of Spinal Anesthesia Induced Itching in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soliman Fakeeh Hospital (Other)
Responsible Party: Principal Investigator, Dr. Amr Aly Ismail Keera, Prof. Amr Aly Keera, Dr. Soliman Fakeeh Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02/IRB/2016
Record Dates: First submitted 2016-10-19; First posted 2016-11-01 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Itching
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (R) Rapid spinal fentanyl injection (Active Comparator): Patients will receive 25 mic fentanyl spinal ( after dilution with 2.5 ml CSF) in 15 seconds then 10 mg hyperbaric bupivacaine.
  Interventions: Drug: (R) Rapid spinal fentanyl injection
- (S) Slow spinal fentanyl injection (Active Comparator): Patients will receive 25 mic fentanyl spinal ( after dilution with 2.5 ml CSF) in 90 seconds then 10 mg hyperbaric bupivacaine.
  Interventions: Drug: (S) Slow spinal fentanyl injection

INTERVENTIONS:
Drug: (R) Rapid spinal fentanyl injection — Patients will receive 25 micrograms fentanyl ( after dilution with 2.5 ml CSF) in 20 seconds then 10 mg hyperbaric bupivacaine.
  Arms: (R) Rapid spinal fentanyl injection
Drug: (S) Slow spinal fentanyl injection — Patients will receive 25 micrograms fentanyl ( after dilution with 2.5 ml CSF) in 90 seconds then 10 mg hyperbaric bupivacaine.
  Arms: (S) Slow spinal fentanyl injection

SUMMARY:
Pruritus is a troublesome side-effect of neuraxial (epidural and intrathecal) opioids. Sometimes it may be more unpleasant than pain itself. The incidence of pruritus is 83% in postpartum patients and 69% in non-pregnant patients including males and females (1). Some researchers concluded that slow injection rate of hyperbaric bupivacaine may be a simple and effective way to reduce the incidence and severity of hypotension during cesarean section under spinal anesthesia (2). In this new research I want to investigate the effect of slow injection of fentanyl separately, in spinal anesthesia for cesarean section, on the incidence of itching In this double blind randomized study two hundred parturient will be randomly allocated in to two groups; Group (R) will receive 25 mic fentanyl spinal ( after dilution with 2.5 ml CSF) in 15 seconds. Group (S) will receive the same dose in 90 seconds All parturient will receive 10 mg bupivacaine in 45 min after fentanyl. Exclusion criteria will be those with allergy to any medications, contraindications to spinal anesthesia, those who requested sedation, presence of skin lesions that may cause itching and opioid addiction.

Parturient will be monitored regarding the incidence of itching, hypotension, nausea and vomiting. Onset and level of sensory block will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective and emergency cesarean section parturient.

Exclusion Criteria:

* Allergy to any medications, contraindications to spinal anesthesia, those who requested sedation, presence of skin lesions that may cause itching and opioid addiction.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
( 0 - 10) Itching scale | 60 min

SECONDARY OUTCOMES:
Satisfactory Block ( no pain, Pain relieved by opioids or pain needs general anesthesia | 60 min

OTHER OUTCOMES:
Hypotension ( yes or no) | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Keera, Principal Investigator — Doctor Soliman Fakeeh Hospital

IPD SHARING:
Plan to Share IPD: Yes
I hope to publish the data in a respected journal.